CLINICAL TRIAL: NCT05506709
Title: A Clinical Research Trial Confirming the Safety and Performance of a Seawater-based Nasal Spray for Relief of Allergic Rhinitis Symptoms
Brief Title: Sterimar Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-20-F12
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Masking Description: Product-blinded (the brand name of the product is not available for subjects)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test (Experimental): Subjects receive only the test product (medical device/nasal pump containing moderately hypertonic solution produced based on 100% natural sea water rich of marine trace elements with added manganese and calcium)
  Interventions: Device: Seawater nasal spray

INTERVENTIONS:
Device: Seawater nasal spray — Subjects will use the nasal spray (moderately hypertonic solution based on 100% natural sea water rich of marine trace elements with added manganese and calcium) at least once and up to 6 times as necessary per day during the 14-day test period. Each application is composed of two irrigating sprays per nostril for a total of 4 sprays per application.

SUMMARY:
The study aims to confirm the safety and performance of a hypertonic seawater-based nasal spray enriched with manganese and calcium, in relief/reduction of nasal symptoms (congestion, itchy nose, runny nose and sneezing) among subjects with symptomatic allergic rhinitis. This will be a prospective, longitudinal, single-cell and product blinded clinical trial. A sufficient number (65-70) of adult subjects with allergic rhinitis meeting all eligibility criteria will be enrolled in this study to ensure that approximately 50 subjects complete the study. Subjects will be enrolled during allergy season. The study will consist of four visits with a total duration of 3 weeks (1 week of pre-screening and 2 weeks for investigational product use). The full schedule of events is presented in the CIP. Subjects recruited for this study will be screened for inclusion/exclusion criteria after reading and signing the informed consent form. Eligible subjects who show a positive reaction to the skin prick test at Visit 1/ Day -7 will be enrolled for a one-week pre-run screening period. At baseline (Visit 2/Day 0), those subjects meeting all inclusion criteria including the results of the Total Nasal Symptoms Score will be enrolled in the active study phase. The subjects will use the product during two weeks (from Day 7 to Day 14), applying at least once and maximum 6 times daily per instructions for use.

At each visit within intervention period (Visits 2, 3 and 4), the subjects will be asked to assess their nasal and ocular symptoms (using Nasal Symptom Score and Ocular Symptom Score grading tools) before product application, as well as at 1 minute, 10 minutes and 1-hour post-product application. Besides, they will complete Weekly Rhinitis questionnaire for the past week. Additionally, the subjects will complete Daily Diaries to record their nasal and ocular symptoms, sleep disturbance, and need for use of other medication.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years of age.
2. Male or female.
3. Self-reported or medical history of allergic rhinitis during the past 18 months.
4. Having a positive skin puncture test (wheal diameter at least 3 mm greater than saline negative control) to at least one pollen of trees, weeds, and grasses meadows. Specific strains will be noted in the skin prick test report [Note: Subjects should also receive skin prick/puncture tests for perennial allergens, and they can be polysensitized to perennial allergens (dust mites, house dust, dog dander, cat dander, feather)].
5. Willingness NOT to use any medications for relief of allergic rhinitis symptoms during the 3 weeks of the study.
6. Being able to read and sign informed consent, as well as fill assessment questionnaire.
7. Daily TNSS ≥6 of possible maximum 12 on at least 3 consecutive days, or daily TNSS ≥5 of possible maximum of 12 with one symptom being severe on at least 3 consecutive days of the 1-week run-in period before the baseline visit (Visit 2/Day 0) (based on the nasal symptoms listed in Appendix I). Daily TNSS is the average of morning (within 15 minutes of awakening) and evening TNSS (within an hour before going to bed) to be calculated by the study staff at baseline (Visit 2/Day 0)

Exclusion Criteria:

1. Any symptoms of upper or lower respiratory tract infections within 2 weeks prior to the first visit or during the study.
2. Positive COVID -19 test during the past month or during the course of the study.
3. Self-reported history of anaphylaxis.
4. Confirmed diagnosis of urticaria or eczema.
5. Confirmed diagnosis of asthma that requires more than intermittent rescue beta agonist treatment, for example, prior to exercise.
6. Immunotherapy during the past 2 years, or ongoing immunotherapy.
7. Recent nasal or sinus surgery within the last 6 months.
8. Use of any OTC and prescription antihistamine, cromone, decongestant, systemic/topical corticosteroids, leukotriene antagonists, topical antibiotics, non-steroidal anti-inflammatory drugs in the past 2 weeks.
9. Use of other nasal sprays, pump, CPAP machine, nasal irrigation/lavage devices, internal nasal gel or nasal oil within 2 weeks prior to the first visit or during the study.
10. Women who are pregnant and/or breastfeeding or planning to become pregnant during the study and within 30 days after the last application of the study product.
11. Presence of nasal polyposis, chronic sinusitis (assessed by Investigator).
12. Nasal anatomic abnormality (assessed by Investigator), e.g., severe deviated septum, congenital cleft lip/palate, nasal bleeding diathesis.
13. Any clinically significant co-morbid condition, which, in PI's opinion, may affect the patient safety and/or affect participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | Through study completion, an average of 3 weeks
  The Total Nasal Symptom Score (TNSS) is the sum of the 4 individual nasal symptoms scores: nasal itching, congestion, runny nose, sneezing. Symptoms will be assessed by questionnaire with scoring from 0 (none) to 3(severe).
Nasal Symptom Score (NSS) for (congestion (stuffy/blocked nose) | Through study completion, an average of 3 weeks
  Nasal Symptom Score (NSS) will be assessed by questionnaire with scoring from 0 (none) to 3(severe).
Nasal Symptom Score (NSS) for sneezing | Through study completion, an average of 3 weeks
  Nasal Symptom Score (NSS) will be assessed by questionnaire with scoring from 0 (none) to 3(severe).
Nasal Symptom Score (NSS) for itching | Through study completion, an average of 3 weeks
  Nasal Symptom Score (NSS) will be assessed by questionnaire with scoring from 0 (none) to 3(severe).
Nasal Symptom Score (NSS) for runny nose | Through study completion, an average of 3 weeks
  Nasal Symptom Score (NSS) will be assessed by questionnaire with scoring from 0 (none) to 3(severe).

SECONDARY OUTCOMES:
Total Ocular Symptom Score (TOSS) | Through study completion, an average of 3 weeks
  The Total Ocular Symptom Score (TOSS) comprised of the sum of the 4 individual ocular symptoms scores: itching, watering, puffy eyes, dry/irritated/burning eyes.
Ocular Symptom Score (OSS) for itching | Through study completion, an average of 3 weeks
  Ocular Symptom Score (OSS) will be assessed by questionnaire with scoring from 0 (none) to 3(severe).
Ocular Symptom Score (OSS) for watering | Through study completion, an average of 3 weeks
  Ocular Symptom Score (OSS) will be assessed by questionnaire with scoring from 0 (none) to 3(severe).
Ocular Symptom Score (OSS) for puffy eyes | Through study completion, an average of 3 weeks
  Ocular Symptom Score (OSS) will be assessed by questionnaire with scoring from 0 (none) to 3(severe).
Ocular Symptom Score (OSS) for dry/irritated/burning eyes | Through study completion, an average of 3 weeks
  Ocular Symptom Score (OSS) will be assessed by questionnaire with scoring from 0 (none) to 3(severe).
Onset of relief (immediate relief) | Through study completion, an average of 3 weeks
  Onset of relief will be using TNSS and individual NSS scores assessed at 1min, 10min and 1 hour after product application.
Duration of relief (long-lasting) | Through study completion, an average of 3 weeks
  Duration of relief using the time between first and second daily applications. Time of application will be recorded by subject daily.

OTHER OUTCOMES:
Weekly Rhinitis Control | Through study completion, an average of 3 weeks
  Subjects will complete Weekly rhinitis control questionnaire for the past week. They grade their symptoms during the week from 5 to 1, where higher score means better outcome
Need of other medications | Through study completion, an average of 3 weeks
  subjects will be asked whether they need other medication to treat their symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- "Heratsi" Hospital Complex No.1, Yerevan, Armenia